CLINICAL TRIAL: NCT04654130
Title: An Effectiveness Trial Examining Neurofeedback in Adults With PTSD
Brief Title: Neurofeedback Effectiveness Trial in PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to challenges with the COVID-19 pandemic, our team has had to prioritize certain studies, which means we can no longer pursue this study at our site.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: McMaster University (Other); FDC Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10500; 116730 (Other: Western University's Research Ethics Board)
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-03

CONDITIONS: PTSD; Post-traumatic Stress Disorder; Cognitive Dysfunction; Cognitive Deficit
Keywords: neurofeedback; ICN; intrinsic connectivity networks; default mode network; salience network
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Cognitive Dysfunction; Cognition Disorders | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: This study is an effectiveness trial investigating neurofeedback as an intervention for both symptoms of PTSD, and the commonly associated cognitive impairment/dysfunction (e.g., attention, executive function, processing speed). Participants will be randomized to one of two conditions: NFB or Wait List.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback (NFB) (Experimental): Participants in the NFB condition will complete 19 weekly sessions of NFB from home with research staff supervision (via videoconferencing), and pre-, post- and 3-month follow-up assessments.
  Interventions: Other: Neurofeedback
- Wait List (No Intervention): Participants in the Wait List condition will receive no NFB for approximately 31 weeks, and will be asked to complete pre-, post- and 3-month follow-up assessments. After study completion, they will be offered the same 19 weeks of NFB.

INTERVENTIONS:
Other: Neurofeedback — NFB is a type of brain training in which a person is given real-time information (or feedback) from their own brain activities to help them potentially change how their brain is functioning (i.e., to work in a healthier or more effective manner). In the current study, we will implement at-home, supervised (via teleconferencing) neurofeedback sessions using the Muse headband paired with the Myndlift software application to conduct "alpha-down" neurofeedback once per week, for 19 weeks.
  Other Names: EEG Biofeedback
  Arms: Neurofeedback (NFB)

SUMMARY:
This study is an effectiveness trial investigating neurofeedback (NFB) in adults with PTSD (Post-Traumatic Stress Disorder). Participants will be randomly assigned to one of two treatment conditions - i) NFB, or ii) wait list. Due to the coronavirus pandemic, our study will, primarily, take place online (i.e., online assessment and treatment, with option of in-person fMRI, or functional magnetic resonance imaging, scans). NFB sessions will be conducted from home, with videoconferenced supervision by research staff. After study completion, individuals in the wait list condition will be offered the same NFB treatment.

DETAILED DESCRIPTION:
PTSD has an emotional impact on individuals, but it is also associated with impaired cognitive functioning (e.g., processing speed, attention, executive functioning). Unfortunately, there is little research investigating both issues simultaneously. The current study is an effectiveness trial for an intervention called neurofeedback (NFB), which may be helpful in addressing both PTSD symptom severity, and cognitive dysfunction. NFB is a type of brain training in which a person is given real-time information (or feedback) from their own brain activity to help them potentially change how their brain is functioning (i.e., to work in a healthier or more effective manner). NFB has been in use for over 30 years, and it is proven to be quite effective in treating ADHD (Attention Deficit Hyperactivity Disorder); however, it has not been embraced as a clinical intervention for other mental health disorders. Recent systematic reviews of NFB suggest that this treatment intervention can lead to significant clinical improvements (e.g., reduction in PTSD severity), and it can impact both functional brain activity and cognitive function. The current study hopes to bring these 3 areas of interest together by investigating the impact of NFB on PTSD symptoms, cognitive ability, and intrinsic neurological connectivity (via fMRI - function magnetic imaging).

In the current study, participants will be randomized into one of two conditions: NFB or Wait List. Those in the NFB condition will begin 19 weekly, supervised (via teleconferencing) sessions of NFB, while the Wait List will not receive NFB for approximately 31 weeks (i.e., not until final assessments are complete). After all assessments are complete, participants in the Wait List condition will be able to begin the same 19 sessions of NFB. Study participation includes pre-, post-, and 3-month follow-up assessments, and 2 optional fMRI scans. Due to the current coronavirus pandemic, this study will be conducted primarily online.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of PTSD as determined by our pre-treatment assessment
* Due to online nature: must have access to (and ability to use) a computer/tablet with a working microphone and camera (or webcam) for assessments, and a tablet/smartphone for NFB, reliable access to a secure internet connection, and access to a quiet, private space for the assessments and sessions.
* Ability to provide informed consent
* Fluency in written and spoken English
* must be resident of Ontario (due to restrictions of professional licenses)

Exclusion Criteria for those opting in to fMRI scan:

* any implants, conditions, etc. that do not comply with 7T (Tesla) fMRI research safety standards (e.g., pacemaker, pregnancy/possible pregnancy)

Exclusion Criteria for study in general:

* history of significant head injury/lengthy loss of consciousness (e.g., a Glasgow Coma Scale Score < 15 at the time of incident as assessed retrospectively by participant)
* significant untreated medical illness
* history of neurological or neurodevelopmental disorder
* history of any pervasive developmental disorder
* any medical disorder known to adversely affect cognition within the last 12 months
* lifetime bipolar or psychotic disorder
* alcohol/substance abuse or dependence within the last 3 months
* extensive narcotic use (e.g., fentanyl, oxycodone, etc.), use of anti-cholinergics, anti-psychotics, psychostimulants, or benzodiazepines
* ECT (electroconvulsive therapy) within the last 12 months
* significant dissociative disorder (as determined by our baseline assessment)
* suicide attempt in last 6 months
* pregnancy (due to impact of hormones on cognitive abilities)
* hearing or vision issues that would interfere with effective online participation:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale (CAPS) score from baseline to post-treatment assessment. | 19 weeks
  Gold standard, clinician-administered PTSD assessment tool; min. score=0, max.=80, with higher scores representing greater PTSD symptoms
Change in Clinician Administered PTSD Scale (CAPS) score from post-treatment to 3-month follow-up assessment. | 12 weeks
  Gold standard, clinician-administered PTSD assessment tool; min. score=0, max.=80, with higher scores representing greater PTSD symptoms
Change in Sustained Attention to Response Task (SART) scores from baseline to post-treatment assessment | 19 weeks
  A computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target presented amidst a background of frequent non-targets. This task assesses inattentiveness, impulsivity, sustained attention, and vigilance.
Change in Sustained Attention to Response Task (SART) scores from post-treatment to 3-month follow-up assessment | 12 weeks
  A computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target presented amidst a background of frequent non-targets. This task assesses inattentiveness, impulsivity, sustained attention, and vigilance.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Lanius, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only coded data will be shared with co-investigators who are registered with the study's ethics board application.

REFERENCES:
- [Background] Kluetsch RC, Ros T, Theberge J, Frewen PA, Calhoun VD, Schmahl C, Jetly R, Lanius RA. Plastic modulation of PTSD resting-state networks and subjective wellbeing by EEG neurofeedback. Acta Psychiatr Scand. 2014 Aug;130(2):123-36. doi: 10.1111/acps.12229. Epub 2013 Nov 25. PMID 24266644
- [Background] Rogel A, Loomis AM, Hamlin E, Hodgdon H, Spinazzola J, van der Kolk B. The impact of neurofeedback training on children with developmental trauma: A randomized controlled study. Psychol Trauma. 2020 Nov;12(8):918-929. doi: 10.1037/tra0000648. Epub 2020 Jul 13. PMID 32658503
- [Background] Nicholson AA, Ros T, Densmore M, Frewen PA, Neufeld RWJ, Theberge J, Jetly R, Lanius RA. A randomized, controlled trial of alpha-rhythm EEG neurofeedback in posttraumatic stress disorder: A preliminary investigation showing evidence of decreased PTSD symptoms and restored default mode and salience network connectivity using fMRI. Neuroimage Clin. 2020;28:102490. doi: 10.1016/j.nicl.2020.102490. Epub 2020 Nov 5. PMID 33395981
- [Background] Nicholson AA, Rabellino D, Densmore M, Frewen PA, Paret C, Kluetsch R, Schmahl C, Theberge J, Ros T, Neufeld RWJ, McKinnon MC, Reiss JP, Jetly R, Lanius RA. Intrinsic connectivity network dynamics in PTSD during amygdala downregulation using real-time fMRI neurofeedback: A preliminary analysis. Hum Brain Mapp. 2018 Nov;39(11):4258-4275. doi: 10.1002/hbm.24244. Epub 2018 Jul 13. PMID 30004602